CLINICAL TRIAL: NCT04140344
Title: The NOTICE Study: Neurosurgery and OrThopedIcs Communication Evaluation Study Following Lumbar Fusions
Acronym: NOTICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00103904
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Spine Degeneration; Lumbar Spine Instability; Lumbar Spondylosis
Keywords: Lumbar Fusion; Text Message
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Intervention Model Description: Following baseline assessments, subjects will be randomized with equal probability to one of two arms: 1). The experimental arm, which will receive automated standardized text messages at predetermined intervals, occurring daily the first week post-operatively and gradually tapering over the second week; 2). The control arm - where subjects will not receive any scheduled contact (outside of standard of care phone interactions). All subjects will receive a phone call 30 days (up to 37 days) post-discharge in order to complete the study questionnaires.
Who Masked: Participant
Masking Description: Participants will be told they will receive appropriate information about their spine surgery (including instructions on proper wound care, mobility, and signs and symptoms of infection) in general, either through phone calls, text messages and/or handouts, without specifying the difference between the control and the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1: Text Message Group (Experimental): The intervention group will receive automated text messages every day for the first week, and every other day for the second week post-operatively. The text messages will follow a series of pre-defined standardized scripts (Appendix 3) with embedded hyperlinks to a video from the providers with further advice. The patient is directed not to respond to the text messages, but to call for any questions or concerns. The text message group will receive a 30-day post-operative phone call to evaluate: number of ED visits, hospital readmissions, and to re-administer the questionnaires completed at baseline visit. Other data to be collected may include the following: number of phone calls to provider, MyChart messages to provider, pain medications, and new problems like pain and infection.
  Interventions: Other: Text Message Group
- ARM 2: Control group (No Intervention): The control group will be given the standard post-op packet that includes detailed instructions on proper wound care and signs and symptoms of infection. They will not receive text messages. The same outcomes will be assessed in both groups through a 30-day post-operative phone call.

INTERVENTIONS:
Other: Text Message Group — The intervention group will receive automated text messages every day for the first week, and every other day for the second week post-operatively. The text messages will follow a series of pre-defined standardized scripts (Appendix 3) with embedded hyperlinks to a video from the providers with further advice. The patient is directed not to respond to the text messages, but to call for any questions or concerns. The text message group will receive a 30-day post-operative phone call to evaluate: number of ED visits, hospital readmissions, and to re-administer the questionnaires completed at baseline visit. Other data to be collected may include the following: number of phone calls to provider, MyChart messages to provider, pain medications, and new problems like pain and infection.
  Other Names: Guidance via text messaging to lumbar spine surgery patients post-operatively
  Arms: ARM 1: Text Message Group

SUMMARY:
The purpose of this single-blind, randomized, controlled study is to assess the efficacy of "informative text messages" vs "traditional handouts" provided to lumbar spine surgery patients post-operatively.

DETAILED DESCRIPTION:
A total of 224 adult patients (18 years or older) undergoing spinal fusion surgery at Duke University Hospital, will be recruited from the Duke Department of Neurosurgery and the Duke Department of Orthopedics. Participants will be consented and will complete standard of care outcomes questionnaires (Visual Analogue Scale, Oswestry Disability Index and Euro-Quol 5D) at the pre-operative clinic visit for baseline comparison. Participants will be randomized, through REDCap, with equal probability to either: A) the control group, with standard post-surgery handouts, or B) the experimental group, which will receive text messages for a period of 2 weeks after surgery (daily for the first week, and every other day for the second week). Text messages were designed to be standardized and automated, with an embedded link to a video regarding at-home, post-surgery-care instructions. Patients will be directed not to respond to the text messages, but to call for any questions or concerns. The primary outcome will be a reduction in 30-days post-surgery readmission rates. The secondary outcomes will be a reduction in 30-days post-surgery ED visits rates, back and leg pain scores, and anxiety levels. These outcomes will be assessed via a phone interview at 30-days (up to max of 37 days) post-discharge for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Primary lumbar fusion 1-4 levels
2. 18 years or older
3. Degenerative spine diagnosis
4. Answers YES to all the following screening questions:

   * Do you own a mobile phone that is capable of sending and receiving text messages?
   * Do you know how to text and feel comfortable texting?
   * Are you a regular (at least once a day) text-message user?
   * Are you agreeable to regular contact?

Exclusion Criteria:

1. Prior lumbar fusions
2. Tumors/infection/trauma
3. Prisoners or institutionalized patients
4. Non-English speaking patients
5. Patients who smokes or with uncontrolled diabetes
6. Participants will be removed from study if discharged to a rehabilitation center or discharged beyond 7 days post-operatively (we are expecting ~15% of patients to be discharged to a rehabilitation center or discharged beyond 7 days post-operatively)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in readmission rates within 30 days post-lumbar spine surgery. | Baseline, 30 days
  Change in readmission rates within 30 days post-lumbar spine surgery as measured by questionnaire.

SECONDARY OUTCOMES:
Change in Emergency Department (ED) visit rates within 30 days post-lumbar spine surgery. | Baseline, 30 days
  Change in Emergency Department (ED) visit rates within 30 days post-lumbar spine surgery as measured by questionnaire.
Change in back and leg pain levels within 30 days post-lumbar spine surgery as measured by "Oswestry Disability Index" (ODI) questionnaire. | Baseline, 30 days
  ODI questionnaire is a tool to evaluate a subjective level of functional disability in daily living activities in patients with low back pain. Scores go from 0% (no disability) to 100% (maximum disability possible).
Change in anxiety/depression levels within 30 days post-lumbar spine surgery as measured by "European Quality of Life-5 Dimension" (EQ-5D) questionnaire. | Baseline, 30 days
  The EQ-5D is an instrument to quantify health-related quality of life. Scores can be reported as a five digit number in a range from 11111 (full health) to 55555 (worst health).

OTHER OUTCOMES:
Change in patient satisfaction levels within 30 days post-lumbar spine surgery. | Baseline, 30 days
  Change in patient satisfaction levels within 30 days post-lumbar spine surgery as measured by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Oren N Gottfried, MD FAANS, Principal Investigator — Duke Neurosurgery
Locations (1):
- Duke Neurosurgery and Duke Orthopedics, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No